CLINICAL TRIAL: NCT07347886
Title: Clinical Outcomes of Sedation in Cataract Surgery Performed Under Topical Anesthesia
Acronym: SADCAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Bekzat Emilbekov, Research Assistant in Anesthesiology, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1503993
Record Dates: First submitted 2025-12-27; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cataract
Keywords: Topical anesthesia, sedation, patient satisfaction, ISAS-T
MeSH Terms: conditions — Cataract; Patient Satisfaction | interventions — Saline Solution; PACEBO protocol; Midazolam; Fentanyl

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three parallel groups, each receiving a different sedation strategy during cataract surgery under topical anesthesia.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants and the operating surgeon will be blinded to group allocation. Study medications, including placebo saline in the non-sedation group, will be prepared in identical syringes by an independent clinician not involved in patient care or outcome assessment. Sedative agents will be administered in equal volumes to maintain blinding. Postoperative outcomes, including patient satisfaction, will be evaluated by a blinded outcome assessor.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Topical anesthesia only (placebo) (Placebo Comparator): Patients will receive topical anesthesia for cataract surgery. An intravenous placebo (normal saline) will be administered in an identical volume to maintain blinding. No sedative or opioid medication will be given.
  Interventions: Drug: Normal Saline
- Topical anesthesia + midazolam (Experimental): Patients will receive topical anesthesia combined with intravenous midazolam administered for sedation during cataract surgery. The medication will be prepared and administered in a standardized dose and volume to maintain blinding.
  Interventions: Drug: Midalozam
- Topical anesthesia + midazolam + fentanyl (Experimental): Patients will receive topical anesthesia combined with intravenous midazolam and fentanyl for sedation during cataract surgery. Medications will be administered in standardized doses and equal volumes to ensure blinding across study groups.
  Interventions: Drug: Midalozam; Drug: Fentanyl (IV)

INTERVENTIONS:
Drug: Normal Saline — Intravenous normal saline administered in an identical volume as placebo to maintain blinding. No sedative or opioid medication will be given.
  Other Names: Pacebo
  Arms: Topical anesthesia only (placebo)
Drug: Midalozam — Intravenous midazolam administered for procedural sedation during cataract surgery performed under topical anesthesia. The medication will be prepared and administered in standardized doses and identical volumes to maintain blinding.
  Other Names: Dormicum
  Arms: Topical anesthesia + midazolam; Topical anesthesia + midazolam + fentanyl
Drug: Fentanyl (IV) — intravenous fentanyl administered in combination with midazolam to provide analgesia and sedation during cataract surgery under topical anesthesia. The medication will be prepared and administered in standardized doses and equal volumes to ensure blinding across study groups.
  Other Names: Fentanyl citrtate
  Arms: Topical anesthesia + midazolam + fentanyl

SUMMARY:
This study aims to evaluate the clinical outcomes of different sedation strategies in patients undergoing cataract surgery performed under topical anesthesia. Cataract surgery is commonly performed under topical anesthesia; however, some patients may experience anxiety, discomfort, or inadequate cooperation during the procedure. Sedation may improve patient comfort and surgical conditions, but it may also be associated with potential adverse effects.

In this randomized, prospective study, patients will be assigned to one of three groups: topical anesthesia alone, topical anesthesia combined with midazolam, or topical anesthesia combined with midazolam and fentanyl. Intraoperative sedation levels, hemodynamic parameters, patient satisfaction, and surgeon satisfaction will be assessed and compared among the groups.

The results of this study are expected to provide evidence regarding the effectiveness and safety of sedation during cataract surgery performed under topical anesthesia and to help optimize perioperative sedation strategies for these patients.

DETAILED DESCRIPTION:
Cataract surgery is one of the most frequently performed ophthalmologic procedures and is commonly carried out under topical anesthesia. Although topical anesthesia provides adequate analgesia, some patients may experience anxiety, discomfort, or difficulty in maintaining cooperation during the procedure. Sedation is frequently used as an adjunct to topical anesthesia to improve patient comfort and surgical conditions; however, concerns remain regarding potential respiratory and hemodynamic adverse effects, particularly in elderly patients.

This prospective, randomized clinical study is designed to evaluate the clinical outcomes of different sedation strategies in patients undergoing cataract surgery performed under topical anesthesia. Adult patients scheduled for elective cataract surgery will be randomly assigned to one of three groups. Group 1 will receive topical anesthesia alone without sedation. Group 2 will receive topical anesthesia combined with intravenous midazolam. Group 3 will receive topical anesthesia combined with intravenous midazolam and fentanyl. Randomization will be performed using a predefined allocation method to ensure balanced group distribution.

All patients will be monitored using standard intraoperative monitoring, including non-invasive blood pressure, electrocardiography, and peripheral oxygen saturation. Supplemental oxygen will be administered when clinically indicated. Sedative agents will be administered according to standardized dosing protocols. Intraoperative sedation depth will be assessed using a validated sedation scale, and hemodynamic and respiratory parameters will be recorded throughout the procedure.

The primary outcome of the study is postoperative patient satisfaction, which will be assessed using the Iowa Satisfaction with Anesthesia Scale - Turkish version (ISAS-T). Secondary outcomes include intraoperative sedation level, surgeon satisfaction, hemodynamic stability, respiratory events, additional sedative requirements, and the occurrence of sedation-related adverse effects. Surgeon satisfaction will be evaluated using a standardized Likert-type scale.

The results of this study are expected to provide evidence regarding the impact of different sedation strategies on patient satisfaction and overall clinical outcomes in cataract surgery performed under topical anesthesia. These findings may contribute to optimizing perioperative sedation practices and improving patient-centered care in ophthalmic anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* American Society of Anesthesiologists (ASA) physical status I-III
* Patients scheduled for elective unilateral cataract surgery
* Surgery planned to be performed under topical anesthesia
* Ability to understand the study procedures and provide written informed consent after being fully informed about the study

Exclusion Criteria:

* Refusal to participate in the study or withdrawal of consent at any stage of the study
* Known intolerance or contraindication to sedative and/or opioid medications
* Presence of significant cardiac arrhythmias
* Severe chronic obstructive pulmonary disease (COPD)
* Hepatic or renal failure
* Inability to cooperate due to cognitive impairment or hearing disability
* Opioid dependence
* Diagnosis of obstructive sleep apnea syndrome (OSAS)
* New York Heart Association (NYHA) class III-IV heart failure
* Conversion to general anesthesia for any reason during surgery

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction after cataract surgery | 1 hour postoperatively
  Patient satisfaction will be assessed using the validated Turkish version of the Iowa Satisfaction with Anesthesia Scale (ISAS-T). The ISAS-T total score will be calculated according to the instrument instructions; higher scores indicate greater satisfaction.

SECONDARY OUTCOMES:
Intraoperative sedation level | During surgery (intraoperative period
  Intraoperative sedation depth will be assessed using the Ramsay Sedation Scale during cataract surgery performed under topical anesthesia.
Preoperative anxiety level | Preoperative period (before surgery)
  Preoperative anxiety will be assessed using the Turkish version of the Amsterdam Preoperative Anxiety and Information Scale (APAIS).
Surgeon satisfaction | Immediately after surgery
  Surgeon satisfaction will be assessed using a 5-point Likert scale.
İntraoperative heart rate | During surgery
  Heart rate will be continuously monitored intraoperatively using standard anesthesia monitoring.
  Values will be recorded at predefined time points during surgery.
İntraoperative mean arterial pressure | During surgery
  Mean arterial pressure will be measured intraoperatively using non-invasive blood pressure monitoring.
  Measurements will be recorded at predefined time points during surgery.
Respiratory events | During surgery
  Intraoperative respiratory events will be assessed using continuous pulse oximetry (SpO₂ monitoring) and clinical airway intervention records.
  Oxygen desaturation will be defined as SpO₂ < 90% lasting ≥ 10 seconds.
  Airway support will be recorded as the need for any of the following interventions: jaw thrust, chin lift, insertion of an oral or nasal airway, or assisted ventilation via face mask.
  Each event will be recorded as a binary outcome (yes/no) during the intraoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Gürcan Güngör, MD, Associate professor, Principal Investigator — İstanbul University-Cerrahpaşa; Cezmi Doğan, MD, Associate professor, Study Chair — İstanbul University-Cerrahpaşa
Locations (1):
- Istanbul University-Cerrahpaşa, Cerrahpaşa Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the nature of this single-center academic thesis study and to protect participant confidentiality. No formal data-sharing agreement has been planned.

REFERENCES:
- [Background] Dexter F, Aker J, Wright WA. Development of a measure of patient satisfaction with monitored anesthesia care: the Iowa Satisfaction with Anesthesia Scale. Anesthesiology. 1997 Oct;87(4):865-73. doi: 10.1097/00000542-199710000-00021. PMID 9357889